CLINICAL TRIAL: NCT02486809
Title: A Phase I, Randomized, Open-Label, Parallel-Group, Single-Dose, Multi-Center Study in Healthy Subjects to Investigate the Bioequivalence Between a High-Concentration Formulation of Lebrikizumab Administered Subcutaneously by a Needle and Syringe and a Low-Concentration Formulation of Lebrikizumab Administered Subcutaneously by a Prefilled Syringe With Needle Safety Device (PFS-NSD)
Brief Title: A Bioequivalence Study of Subcutaneous (SC) Lebrikizumab Administered by Needle and Syringe or by Prefilled Syringe With Needle Safety Device (PFS-NSD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP29651
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — lebrikizumab

ARMS (2):
- Treatment 1: Needle and Syringe (Experimental): Healthy volunteers will receive a single SC injection of lebrikizumab, withdrawn from a vial and administered by a needle and syringe.
  Interventions: Drug: Lebrikizumab
- Treatment 2: PFS-NSD (Experimental): Healthy volunteers will receive a single SC injection of lebrikizumab, administered by PFS-NSD.
  Interventions: Drug: Lebrikizumab

INTERVENTIONS:
Drug: Lebrikizumab — Participants will receive a single SC dose of lebrikizumab, delivered via needle and syringe or PFS-NSD.

SUMMARY:
This study will assess the bioequivalence in healthy participants between a high-concentration formulation of lebrikizumab withdrawn from a vial and administered SC as a single injection by a needle and syringe, and a low-concentration formulation of lebrikizumab administered SC as a single injection via PFS-NSD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18 to 65 years of age, inclusive
* Body mass index (BMI) 18 to 32 kg/m^2 and body weight 50 to 100 kg, inclusive
* Nonpregnant and nonlactating females
* Agreement to utilize effective contraception among men and women of childbearing potential

Exclusion Criteria:

* Known allergy or hypersensitivity to study drug or components
* History of alcohol or drug abuse within 12 months prior to study drug, or positive test for alcohol or drugs of abuse
* Receipt of an investigational agent within 30 days of 5 half-lives prior to Day -1
* Biological therapy within 90 days prior to Day -1
* Parasitic or Listeria monocytogenes infection within 6 months prior to Screening
* Receipt of blood products within 2 months prior to study entry
* Donation or loss of blood/plasma within up to 6 months prior to study drug, depending upon volume
* Receipt of live attenuated vaccine within 1 month prior to study drug
* Use of tobacco- or nicotine-containing products within 14 days prior to Screening
* Use of any prescription or nonprescription medication within 14 days prior to study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of lebrikizumab | Pre-dose and post-dose from Day 1 until study completion or premature withdrawal (up to approximately 3 months)
Time to maximum concentration (Tmax) of lebrikizumab | Pre-dose and post-dose from Day 1 until study completion or premature withdrawal (up to approximately 3 months)
Area under the concentration-time curve to the last measurable concentration (AUC0-last) of lebrikizumab | Pre-dose and post-dose from Day 1 until study completion or premature withdrawal (up to approximately 3 months)
Area under the concentration-time curve extrapolated to infinity (AUC0-inf) of lebrikizumab | Pre-dose and post-dose from Day 1 until study completion or premature withdrawal (up to approximately 3 months)
Apparent terminal elimination rate constant of lebrikizumab | Pre-dose and post-dose from Day 1 until study completion or premature withdrawal (up to approximately 3 months)
Apparent terminal elimination half-life (t1/2) of lebrikizumab | Pre-dose and post-dose from Day 1 until study completion or premature withdrawal (up to approximately 3 months)
Apparent clearance (CL/F) of lebrikizumab | Pre-dose and post-dose from Day 1 until study completion or premature withdrawal (up to approximately 3 months)
Apparent volume of distribution (Vz/F) of lebrikizumab | Pre-dose and post-dose from Day 1 until study completion or premature withdrawal (up to approximately 3 months)

SECONDARY OUTCOMES:
Incidence of adverse events | From Day -1 until study completion or premature withdrawal (up to approximately 3 months)
Incidence of anti-therapeutic antibodies (ATAs) to lebrikizumab | From Day 1 until study completion or premature withdrawal (up to approximately 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Daytona Beach, Florida
  - Evansville, Indiana
  - Dallas, Texas
  - Madison, Wisconsin